CLINICAL TRIAL: NCT00672607
Title: a Clinical Trial to Evaluate the Efficacy and Safety of Agnucaston Tablets in the Treatment of Premenstrual Syndrome (PMS)
Acronym: ACT-RCT-C 01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schwabe-Wenex International Ltd (Industry)
Responsible Party: Helen Guo, Schwabe-Wenex
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Schwabe-Wenex
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Premenstrual Syndrome
Keywords: premenstual syndrome, PMS, clinical trial
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: extracts of Vitex agnus castus tablets
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: extracts of Vitex agnus castus tablets — orally, one tablet daily. Apply for a period of 3 months. Do not interrupt during menses period.
  Other Names: Agnucaston tablets
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To compare the efficacy and safety of Agnucaston tablets with placebo for the treatment of Premenstrual Syndrome (PMS) and assess if Agnucaston tablets are superior to placebo on efficacy or not.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a common disorder in women and consists of somatic and/or behavioral/mood symptoms, which can impair a woman's social and work-related functioning. Some clinical studies with preparations containing Vitex agnus castus have demonstrated a positive effect on PMS with good tolerability. The aim of this clinical trial is to investigate the efficacy and safety of Agnucaston tablets for the therapy of PMS.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of PMS disease
* Age between 18 and 45 years
* Patients is in general good health

Exclusion Criteria:

* Any of the following endocrinological diseases: diabetes mellitus, hypo-/hyperthyreosis, pituitary tumor.
* Clearly kidney or liver disease, abnormal kidney or liver function.
* Any of the following gynecological diseases: endometriosis, mammary carcinoma, intraductal papilloma, galactorrhea, mammary fibroadenoma.
* Prior to the start of the study any planned surgical intervention of the breasts (including cyst puncture), of the uterus and/ or adnexa.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2005-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline (cycle 0) of premenstrual complaints, assessed by the sum score of the 18 items of the PMS-Diary, after 3 cycles under treatment, evaluated for the luteal phase, i.e. the last 7 days prior a menstrual bleeding. | the last 7 days prior a menstrual bleeding

SECONDARY OUTCOMES:
Change from baseline (cycle 0) of the sum score of the 36 questions of the PMTS self-assessment scale after 3 cycles under treatment. | on the 1st-3nd day of menstrual bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China